CLINICAL TRIAL: NCT00683475
Title: A Phase 2, Multicenter, Randomized Study of IMC-A12 or IMC-1121B Plus Mitoxantrone and Prednisone in Metastatic Androgen-Independent Prostate Cancer (AIPC) Following Disease Progression on Docetaxel-Based Chemotherapy
Brief Title: A Study of IMC-A12 or Ramucirumab Plus Mitoxantrone and Prednisone in Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13924; CP18-0601 (Other: ImClone Systems); I4T-IE-JVBS (Other: Eli Lilly and Company)
Record Dates: First submitted 2008-05-19; First posted 2008-05-23 (Estimated); Results first posted 2014-06-18 (Estimated); Last update posted 2014-10-16 (Estimated); Status verified 2014-10

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — cixutumumab; Mitoxantrone; Prednisone; Ramucirumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IMC-1121B (ramucirumab) + Mitoxantrone + Prednisone (Experimental)
  Interventions: Drug: Mitoxantrone; Drug: Prednisone; Biological: IMC-1121B (ramucirumab)
- IMC-A12 + Mitoxantrone + Prednisone (Experimental)
  Interventions: Biological: IMC-A12; Drug: Mitoxantrone; Drug: Prednisone

INTERVENTIONS:
Biological: IMC-A12 — IMC-A12 is to be administered as an I.V. infusion, 6 mg/kg over 1 hour on Days 1, 8, and 15 of each 3-week (21-day) cycle. IMC-A12 treatment is to continue until there is evidence of disease progression, death, intolerable toxicity, or other withdrawal criteria are met.
  Other Names: cixutumumab; LY3012217
  Arms: IMC-A12 + Mitoxantrone + Prednisone
Drug: Mitoxantrone — Mitoxantrone is to be administered as an I.V. infusion, at 12 milligrams/square meter (mg/m^2) over 5-15 minutes on Day 1 during a 3-week (21-day) cycle. Mitoxantrone treatment is to be continued for a maximum of 12 cycles (total cumulative dose of mitoxantrone is restricted to ≤ 144 mg/m^2) or until there is evidence of disease progression, death, or intolerable toxicity.
Drug: Prednisone — Prednisone (5 mg) is to be self-administered PO BID, each day of the 21-day cycle.
Biological: IMC-1121B (ramucirumab) — IMC-1121B (ramucirumab) is to be administered as an intravenous (IV) infusion, 6 milligrams/kilogram (mg/kg) over 1 hour on Days 1, 8, and 15 of each 3-week (21-day) cycle. Ramucirumab treatment is to continue until there is evidence of disease progression, death, intolerable toxicity, or other withdrawal criteria are met.
  Other Names: ramucirumab; IMC-1121B; LY3009806
  Arms: IMC-1121B (ramucirumab) + Mitoxantrone + Prednisone

SUMMARY:
The purpose of this study is to determine whether IMC-A12 or IMC-1121B (ramucirumab) with Mitoxantrone and Prednisone is effective in the treatment of metastatic androgen- independent prostate cancer (APIC).

DETAILED DESCRIPTION:
Prostate cancer is the most frequently diagnosed cancer in men and the second leading cause of cancer-related death in men in the United States. Chemotherapy, either as a single agent or in combination, may lead to clinical response, pain control, and/or improved quality of life. Docetaxel is now the first-line standard therapy for AIPC. Mitoxantrone was approved in 1996 for use in combination with corticosteroids as initial chemotherapy for pain related to advanced Hormone Refractory Prostate Cancer (HRPC). Hormonal manipulations and docetaxel-based chemotherapy are often effective in metastatic prostate cancer; however, disease becomes refractory to these interventions in the majority of men. Although mitoxantrone continues to be a significant agent in the treatment of HRPC, there exists a need for more efficacious therapy in docetaxel-refractory- AIPC. Because of the potential contribution of Insulin Like Growth Factor Receptor (IGF-IR) and VEGFR-2 mediated pathways in prostate cancer pathogenesis, it is hypothesized that each of these biological agents in combination with mitoxantrone and prednisone will result in clinically meaningful activity in AIPC. Therefore, ImClone plans to conduct a randomized Phase 2 trial to assess the safety and efficacy of IMC-A12 or IMC-1121B (ramucirumab) in combination with mitoxantrone and prednisone in participants with AIPC.

ELIGIBILITY:
Inclusion Criteria:

* The participant has histologically-confirmed adenocarcinoma of the prostate
* The participant has radiographic evidence of metastatic prostate cancer (stage M1 or D2)
* The participant has prostate cancer unresponsive or refractory to hormone therapy (androgen-independent)
* The participant has had disease progression (clinical or radiographic) while receiving docetaxel, or within 120 days of receiving docetaxel-based chemotherapy and in the opinion of the investigator is unlikely to derive significant benefit from additional docetaxel-based therapy, or was intolerant to therapy with this agent
* The participant must have evidence of progressive disease defined as at least one of the following;

  1. Progressive measurable disease: using conventional solid tumor criteria
  2. Bone scan progression: at least two new lesions on bone scan
  3. Increasing PSA: at least two consecutive rising PSA values over a reference value (PSA #1) taken at least 1 week apart. A third PSA (PSA #3) is required to be greater than PSA #2; if not, a fourth PSA (PSA #4) is required to be greater than PSA #2
* The participant has a PSA ≥ 2 ng/mL
* The participant has prior surgical or medical castration with a serum testosterone of <50 ng/mL. If the method of castration is luteinizing hormone releasing level hormone (LHRH) agonists, the participant must be willing to continue the use of LHRH agonists during protocol treatment
* The participant has an Eastern Cooperative Oncology Group performance status (ECOG PS) 0-2
* The participant has adequate hematologic function (absolute neutrophil count [ANC]≥1500/uL, hemoglobin ≥9 g/dL, and platelets ≥100,000/uL)
* The participant has adequate hepatic function (bilirubin ≤ 1.5 times the upper limit of normal (ULN), Aspartate Transaminase (AST) and Alanine Transaminase (ALT) ≤ 3 times the ULN, or ≤ 5 times the ULN if liver metastases are present)
* The participant has adequate renal function (creatinine ≤ 1.5 x ULN or calculated creatinine clearance > 40 mL/min)
* The participant's urinary protein is ≤ 1+ on dipstick or routine urinalysis (UA). If urine dipstick or routine analysis indicates ≥ 2+ proteinuria, then a 24-hour urine must be collected and must demonstrate < 1000 mg of protein in 24 hours to allow participation in the study
* The participant has adequate coagulation function (an international normalized ratio [INR] ≤ 1.5 and a Partial Thromboplastin Time [PTT] ≤ 5 seconds above the ULN [unless on oral anticoagulant therapy]). Participants receiving full-dose anticoagulation therapy are eligible provided they meet all other criteria, are on a stable dose of oral anticoagulant or low molecular weight heparin (and if on warfarin have a therapeutic INR between 2 and 3)
* The participant has a fasting serum glucose level of < 160 mg/dL, or below the ULN

Exclusion Criteria:

* The participant has received more than one prior cytotoxic chemotherapy regimen for metastatic disease. (Participants who have had a treatment break followed by a second docetaxel-based regimen with subsequent disease progression are eligible.)
* The participant has received prior therapy with mitoxantrone for advanced prostate cancer (prior adjuvant therapy with mitoxantrone is permitted)
* The participant has a history of symptomatic congestive heart failure or has a pre-study echocardiogram or multigated acquisition (MUGA) scan with left ventricular ejection fraction (LVEF) that is ≥ 10% below the LLN
* The participant has received radiotherapy ≤ 21 days prior to first dose of IMC-A12 or Ramucirumab
* The participant is receiving corticosteroids (dexamethasone, prednisone, or others) at a dose > 5 mg prednisone orally (PO) two times per day (BID) or equivalent. Participants receiving corticosteroids at higher doses may be eligible if their corticosteroid therapy is tapered to study levels (prednisone 5 mg PO BID) prior to first dose of study medication, without concomitant clinical deterioration
* The participant has known or suspected brain or leptomeningeal metastases
* The participant has uncontrolled or poorly controlled hypertension
* The participant has poorly controlled diabetes mellitus. Inclusion Criteria:
* The participant has histologically-confirmed adenocarcinoma of the prostate
* The participant has radiographic evidence of metastatic prostate cancer (stage M1 or D2)
* The participant has prostate cancer unresponsive or refractory to hormone therapy (androgen-independent)
* The participant has had disease progression (clinical or radiographic) while receiving docetaxel, or within 120 days of receiving docetaxel-based chemotherapy and in the opinion of the investigator is unlikely to derive significant benefit from additional docetaxel-based therapy, or was intolerant to therapy with this agent
* The participant must have evidence of progressive disease defined as at least one of the following;

  1. Progressive measurable disease: using conventional solid tumor criteria
  2. Bone scan progression: at least two new lesions on bone scan
  3. Increasing PSA: at least two consecutive rising PSA values over a reference value (PSA #1) taken at least 1 week apart. A third PSA (PSA #3) is required to be greater than PSA #2; if not, a fourth PSA (PSA #4) is required to be greater than PSA #2
* The participant has a PSA ≥ 2 ng/mL
* The participant has prior surgical or medical castration with a serum testosterone of <50 ng/mL. If the method of castration is luteinizing hormone releasing level hormone (LHRH) agonists, the participant must be willing to continue the use of LHRH agonists during protocol treatment
* The participant has an Eastern Cooperative Oncology Group performance status (ECOG PS) 0-2
* The participant has adequate hematologic function (absolute neutrophil count [ANC]≥1500/uL, hemoglobin ≥9 g/dL, and platelets ≥100,000/uL)
* The participant has adequate hepatic function (bilirubin ≤ 1.5 times the upper limit of normal (ULN), aspartate transaminase [AST] and alanine transaminase [ALT]≤ 3 times the ULN, or ≤ 5 times the ULN if liver metastases are present)
* The participant has adequate renal function (creatinine ≤ 1.5 x ULN or calculated creatinine clearance > 40 mL/min)
* The participant's urinary protein is ≤ 1+ on dipstick or routine urinalysis (UA). If urine dipstick or routine analysis indicates ≥ 2+ proteinuria, then a 24-hour urine must be collected and must demonstrate < 1000 mg of protein in 24 hours to allow participation in the study
* The participant has adequate coagulation function (an international normalized ratio [INR] ≤ 1.5 and a partial thromboplastin time [PTT] ≤ 5 seconds above the ULN [unless on oral anticoagulant therapy]). Participants receiving full-dose anticoagulation therapy are eligible provided they meet all other criteria, are on a stable dose of oral anticoagulant or low molecular weight heparin (and if on warfarin have a therapeutic INR between 2 and 3)
* The participant has a fasting serum glucose level of < 160 mg/dL, or below the ULN

Exclusion Criteria:

* The participant has received more than one prior cytotoxic chemotherapy regimen for metastatic disease. (Participants who have had a treatment break followed by a second docetaxel-based regimen with subsequent disease progression are eligible.)
* The participant has received prior therapy with mitoxantrone for advanced prostate cancer (prior adjuvant therapy with mitoxantrone is permitted)
* The participant has a history of symptomatic congestive heart failure or has a pre-study echocardiogram or multigated acquisition (MUGA) scan with left ventricular ejection fraction (LVEF) that is ≥ 10% below the LLN
* The participant has received radiotherapy ≤ 21 days prior to first dose of IMC-A12 or Ramucirumab
* The participant is receiving corticosteroids (dexamethasone, prednisone, or others) at a dose > 5 mg prednisone orally (PO) two times per day (BID) or equivalent. Participants receiving corticosteroids at higher doses may be eligible if their corticosteroid therapy is tapered to study levels (prednisone 5 mg PO BID) prior to first dose of study medication, without concomitant clinical deterioration
* The participant has known or suspected brain or leptomeningeal metastases
* The participant has uncontrolled or poorly controlled hypertension
* The participant has poorly controlled diabetes mellitus. Participants with a history of diabetes are allowed to participate, provided that their blood glucose is within normal range (fasting < 120 mg/dL or below ULN) and that they are on a stable dietary or therapeutic regimen for this condition
* The participant has a known human immunodeficiency virus infection or acquired immunodeficiency syndrome-related illness with a history of diabetes are allowed to participate, provided that their blood glucose is within normal range (fasting < 120 mg/dL or below ULN) and that they are on a stable dietary or therapeutic regimen for this condition
* The participant has a known human immunodeficiency virus infection or acquired immunodeficiency syndrome-related illness

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2008-08; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (31):
- United States (31):
  - ImClone Investigational Site, La Jolla, California
  - ImClone Investigational Site, New Haven, Connecticut
  - ImClone Investigational Site, Boca Raton, Florida
  - ImClone Investigational Site, Port Saint Lucie, Florida
  - ImClone Investigational Site, Atlanta, Georgia
  - ImClone Investigational Site, Chicago, Illinois
  - ImClone Investigational Site, Chlcago, Illinois
  - ImClone Investigational Site, Evanston, Illinois
  - ImClone Investigational Site, Maryville, Illinois
  - ImClone Investigational Site, Cedar Rapids, Iowa
  - ImClone Investigational Site, Metairie, Louisiana
  - ImClone Investigational Site, Ann Arbor, Michigan
  - ImClone Investigational Site, Rochester, Minnesota
  - ImClone Investigational Site, St Louis, Missouri
  - ImClone Investigational Site, Billings, Montana
  - ImClone Investigational Site, Roseland, New Jersey
  - ImClone Investigational Site, Buffalo, New York
  - ImClone Investigational Site, East Setauket, New York
  - ImClone Investigational Site, New York, New York
  - ImClone Investigational Site, Durham, North Carolina
  - ImClone Investigational Site, Cleveland, Ohio
  - ImClone Investigational Site, Philadelphia, Pennsylvania
  - ImClone Investigational Site, Pittsburgh, Pennsylvania
  - ImClone Investigational Site, Greenville, South Carolina
  - ImClone Investigational Site, Knoxville, Tennessee
  - ImClone Investigational Site, Nashville, Tennessee
  - ImClone Investigational Site, Abilene, Texas
  - ImClone Investigational Site, Dallas, Texas
  - ImClone Investigational Site, Houston, Texas
  - ImClone Investigational Site, Seattle, Washington
  - ImClone Investigational Site, Madison, Wisconsin

REFERENCES:
- [Derived] Hussain M, Rathkopf D, Liu G, Armstrong A, Kelly WK, Ferrari A, Hainsworth J, Joshi A, Hozak RR, Yang L, Schwartz JD, Higano CS. A randomised non-comparative phase II trial of cixutumumab (IMC-A12) or ramucirumab (IMC-1121B) plus mitoxantrone and prednisone in men with metastatic docetaxel-pretreated castration-resistant prostate cancer. Eur J Cancer. 2015 Sep;51(13):1714-24. doi: 10.1016/j.ejca.2015.05.019. Epub 2015 Jun 13. PMID 26082390

RESULTS

PARTICIPANT FLOW:
Groups:
- IMC-A12 + Mitoxantrone + Prednisone: IMC-A12 intravenous infusion at 6 milligrams/kilogram (mg/kg) on Days 1, 8, and 15 of each 21-day cycle. Mitoxantrone intravenous infusion at 12 milligrams/square meter (mg/m^2) on Day 1 of each 21-day cycle. Prednisone at 5 milligrams (mg) is to be self-administered orally, each day of the 21-day cycle.
- IMC-1121B (Ramucirumab) + Mitoxantrone + Prednisone: IMC-1121B (ramucirumab) intravenous infusion, 6 milligrams/kilogram (mg/kg) on Days 1, 8, and 15 of each 21-day cycle. Mitoxantrone intravenous infusion at 12 milligrams/square meter (mg/m^2) on Day 1 of each 21-day cycle. Prednisone at 5 milligrams (mg) is to be self-administered orally, each day of the 21-day cycle.
Period: Overall Study
Arm/Group | IMC-A12 + Mitoxantrone + Prednisone | IMC-1121B (Ramucirumab) + Mitoxantrone + Prednisone
Started | 69 | 69
Received Any Quantity of Study Drug | 66 | 66
Completed | 65 | 66
Not Completed | 4 | 3
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Never Treated: Adverse Event | 2 | 3
Not completed — Never Treated: Progressive Disease | 1 | 0

BASELINE CHARACTERISTICS:
Population: Modified intent to treat population (mITT): All participants who received any quantity of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | IMC-A12 + Mitoxantrone + Prednisone | IMC-1121B (Ramucirumab) + Mitoxantrone + Prednisone | Total
Number analyzed (Participants) | 66 | 66 | 132
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 21 | 51
  >=65 years | 36 | 45 | 81
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 66 | 66 | 132
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 65 | 63 | 128
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 61 | 58 | 119
  Black Or African American | 4 | 6 | 10
  Other | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 66 | 66 | 132

OUTCOME MEASURES:

1. Primary Outcome: Composite Progression-free Survival (cPFS)
Description: Defined as the median time from randomization to the earliest of:
  1. Tumor progression by Response Evaluation Criteria in Solid Tumors (RECIST);
  2. Evidence of progression by bone scan, performed after completion of the first 3 cycles, demonstrating the appearance of >=2 new lesions;
  3. New skeletal events (New pathologic bone fracture in the region of metastatic disease; New bone lesion requiring radiation or surgery; Spinal cord or nerve root compression)
  4. Symptomatic progression (for participants without measurable disease);
  5. Other clinical events attributable to prostate cancer that require major interventions; or
  6. Death from any cause
  Participants who were ongoing with no progression or who discontinued treatment for reasons other than progression were censored at date of last assessment. Participants who started new anticancer treatment before progression were censored at date of last assessment before start of new anti-cancer therapy.
Time Frame: Randomization to composite progressive disease, up to 23.4 months
Population: Modified intent to treat population (mITT): All participants who received any quantity of study drug.
  11 participants were censored in the IMC-A12 + Mitoxantrone + Prednisone arm. 15 participants were censored in the IMC-1121B (ramucirumab) + Mitoxantrone + Prednisone arm.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | IMC-A12 + Mitoxantrone + Prednisone | IMC-1121B (Ramucirumab) + Mitoxantrone + Prednisone
Number analyzed (Participants) | 66 | 66
months | 4.1 [2.2 to 5.6] | 6.7 [4.5 to 8.3]

2. Secondary Outcome: Summary Listing of Participants Reporting Treatment-Emergent Adverse Events
Description: Data presented are the number of participants who experienced A12 or 1121B (ramucirumab) related treatment-emergent adverse events (TEAE), treatment related serious adverse events (SAE), or any Grade 3 or higher TEAE; any TEAE leading to discontinuation of A12 or 1121B (ramucirumab) treatment, and any TEAE leading to dose modification of A12 or 1121B (ramucirumab). A summary of SAEs and other nonserious AEs, regardless of causality, is located in the Reported Adverse Event section.
Time Frame: Randomization to 36.3 months
Population: Modified intent to treat population (mITT): All participants who received any quantity of study drug.
Measure: Number; unit: participants
Arm/Group | IMC-A12 + Mitoxantrone + Prednisone | IMC-1121B (Ramucirumab) + Mitoxantrone + Prednisone
Number analyzed (Participants) | 66 | 66
participants
  A12/1121B Related TEAE | 64 | 63
  A12/1121B Related Serious TEAE | 22 | 16
  A12/1121B Related Grade >= 3 TEAE | 35 | 31
  TEAE Leading to Dose Modification of A12/1121B | 35 | 35
  TEAE Leading to Discontinuation of A12/1121B | 18 | 25

3. Secondary Outcome: Time to Radiographic Evidence of Disease Progression
Description: Time between date of randomization and earliest date of radiographic progression defined as either:
  1. Tumor progression by RECIST;
  2. Evidence of progression by bone scan;
  3. New skeletal events (New pathologic bone fracture in the region of metastatic disease; New bone lesion requiring radiation or surgery; Spinal cord or nerve root compression).
  Participants who were ongoing with no radiographic evidence of disease progression, who discontinued treatment for reasons other than progression,or died before progression were censored at date of last tumor or bone radiographic assessment. Participants who started a new anticancer treatment before progression were censored at date of last tumor or bone radiographic assessment before start of new anti-cancer therapy.
Time Frame: Randomization to date of radiographic progression, up to 36.3 months
Population: Modified intent to treat population (mITT): All participants who received any quantity of study drug.
  34 participants were censored in IMC-A12 arm and 34 participants were censored in IMC-1121B (ramucirumab) arm.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | IMC-A12 + Mitoxantrone + Prednisone | IMC-1121B (Ramucirumab) + Mitoxantrone + Prednisone
Number analyzed (Participants) | 66 | 66
months | 7.5 [4.8 to 10.1] | 10.2 [7.5 to 12.6]

4. Secondary Outcome: Prostate Specific Antigen (PSA) Response Rate
Description: PSA response rate is defined as the percentage of participants with a decrease in PSA >= 50 percent from baseline.
Time Frame: Baseline up to data cut-off date (up to 36.3 months)
Population: Participants who received any quantity of study drug, had baseline PSA value >= 2 ng/ml and at least one non-missing post-baseline PSA.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IMC-A12 + Mitoxantrone + Prednisone | IMC-1121B (Ramucirumab) + Mitoxantrone + Prednisone
Number analyzed (Participants) | 54 | 56
percentage of participants | 18.5 [9.3 to 31.4] | 21.4 [11.6 to 34.4]

5. Secondary Outcome: Composite Progression-free Survival (cPFS) at 6-months
Description: Data presented are the percentage of participants without disease progression at 6 months.
  Participants who were ongoing with no progression or who discontinued treatment for reasons other than progression were censored at date of last assessment. Participants who started new anticancer treatment before progression were censored at date of last assessment before start of new anti-cancer therapy.
Time Frame: 6 months
Population: Modified intent to treat population (mITT): All participants who received any quantity of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IMC-A12 + Mitoxantrone + Prednisone | IMC-1121B (Ramucirumab) + Mitoxantrone + Prednisone
Number analyzed (Participants) | 66 | 66
percentage of participants | 37.2 [25.0 to 49.4] | 59.2 [45.8 to 70.4]

6. Secondary Outcome: Composite Progression-free Survival (cPFS) at 9-months
Description: Data presented are the percentage of participants without disease progression at 9 months.
  Participants who were ongoing with no progression or who discontinued treatment for reasons other than progression were censored at date of last assessment. Participants who started new anticancer treatment before progression were censored at date of last assessment before start of new anti-cancer therapy.
Time Frame: 9 months
Population: Modified intent to treat population (mITT): All participants who received any quantity of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IMC-A12 + Mitoxantrone + Prednisone | IMC-1121B (Ramucirumab) + Mitoxantrone + Prednisone
Number analyzed (Participants) | 66 | 66
percentage of participants | 20.7 [11.2 to 32.1] | 35.9 [23.4 to 48.5]

7. Secondary Outcome: Composite Progression-free Survival (cPFS) at 12-months
Description: Data presented are the percentage of participants without disease progression at 12 months.
  Participants who were ongoing with no progression or who discontinued treatment for reasons other than progression were censored at date of last assessment. Participants who started new anticancer treatment before progression were censored at date of last assessment before start of new anti-cancer therapy.
Time Frame: 12 months
Population: Modified intent to treat population (mITT): All participants who received any quantity of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IMC-A12 + Mitoxantrone + Prednisone | IMC-1121B (Ramucirumab) + Mitoxantrone + Prednisone
Number analyzed (Participants) | 66 | 66
percentage of participants | 12.4 [5.2 to 22.9] | 20.0 [10.1 to 32.3]

8. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the time from randomization to the date of death due to any cause. Participants who were alive at the time of study completion were censored at the time the participant was last known to be alive.
Time Frame: First dose to death due to any cause up to 36.3 months
Population: Modified intent to treat population (mITT): All participants who received any quantity of study drug.
  Nine participants were censored in the IMC-A12 + Mitoxantrone + Prednisone arm. Twelve participants were censored in the IMC-1121B + Mitoxantrone + Prednisone arm
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | IMC-A12 + Mitoxantrone + Prednisone | IMC-1121B (Ramucirumab) + Mitoxantrone + Prednisone
Number analyzed (Participants) | 66 | 66
months | 10.8 [6.5 to 13.0] | 13.0 [9.5 to 16.0]

9. Secondary Outcome: Objective Response Rate (ORR)
Description: Objective response is Complete Response (CR) + Partial Response (PR), as classified by the investigators according to the Response Evaluation Criteria In Solid Tumors (RECIST) guidelines. CR is a disappearance of all target and non-target lesions; PR is at least a 30% decrease in the sum of the longest diameter of target lesions without new lesions and progression of non-target lesions.
  Objective response rate is calculated as a total number of participants with CR or PR divided by the total number of participants with measurable disease, multiplied by 100.
Time Frame: Baseline to date of progressive disease or death up to 36.3 months
Population: Participants with measurable disease at baseline, who received any quantity of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IMC-A12 + Mitoxantrone + Prednisone | IMC-1121B (Ramucirumab) + Mitoxantrone + Prednisone
Number analyzed (Participants) | 46 | 38
percentage of participants | 15.2 [6.3 to 28.9] | 31.6 [17.5 to 48.7]

10. Secondary Outcome: Maximum Concentration (Cmax) at Study Day 1
Description: Maximum Concentration (Cmax) of Ramucirumab.
  All samples were assayed 36 months post sample collection, which exceeds the established long-term serum stability period for ramucirumab. Therefore, concentration data were invalid and pharmacokinetic (PK) analyses could not be conducted.
Time Frame: Day 1
Population: Zero participants were analyzed.
Groups:
- IMC-1121B (Ramucirumab) + Mitoxantrone + Prednisone: IMC-1121B (ramucirumab) intravenous infusion, 6 milligrams/kilogram (mg/kg) on Days 1, 8, and 15 of each 21-day cycle. Mitoxantrone intravenous infusion at 12 milligrams/square meter (mg/m2) on Day 1 of each 21-day cycle. Prednisone at 5 milligrams (mg) is to be self-administered orally, each day of the 21-day cycle.
Arm/Group | IMC-1121B (Ramucirumab) + Mitoxantrone + Prednisone
Number analyzed (Participants) | 0

11. Secondary Outcome: Maximum Concentration (Cmax) at Study Day 15
Description: as for outcome 10
Time Frame: Day 15
Population: Zero participants were analyzed.
Arm/Group | IMC-1121B (Ramucirumab) + Mitoxantrone + Prednisone
Number analyzed (Participants) | 0

12. Secondary Outcome: Maximum Concentration (Cmax) at Study Day 16
Description: as for outcome 10
Time Frame: Day 16
Population: Zero participants were analyzed.
Arm/Group | IMC-1121B (Ramucirumab) + Mitoxantrone + Prednisone
Number analyzed (Participants) | 0

13. Secondary Outcome: Maximum Concentration (Cmax) at Study Day 30
Description: as for outcome 10
Time Frame: Day 30
Population: Zero participants were analyzed.
Arm/Group | IMC-1121B (Ramucirumab) + Mitoxantrone + Prednisone
Number analyzed (Participants) | 0

14. Secondary Outcome: Minimum Concentration (Cmin) at Study Day 1
Description: Minimum concentration (Cmin) of Ramucirumab.
  All samples were assayed 36 months post sample collection, which exceeds the established long-term serum stability period for ramucirumab. Therefore, concentration data were invalid and pharmacokinetic (PK) analyses could not be conducted.
Time Frame: Day 1
Population: Zero participants were analyzed.
Arm/Group | IMC-1121B (Ramucirumab) + Mitoxantrone + Prednisone
Number analyzed (Participants) | 0

15. Secondary Outcome: Minimum Concentration (Cmin) at Study Day 15
Description: as for outcome 14
Time Frame: Day 15
Population: Zero participants were analyzed.
Arm/Group | IMC-1121B (Ramucirumab) + Mitoxantrone + Prednisone
Number analyzed (Participants) | 0

16. Secondary Outcome: Minimum Concentration (Cmin) at Study Day 16
Description: as for outcome 14
Time Frame: Day 16
Population: Zero participants were analyzed.
Arm/Group | IMC-1121B (Ramucirumab) + Mitoxantrone + Prednisone
Number analyzed (Participants) | 0

17. Secondary Outcome: Minimum Concentration (Cmin) at Study Day 30
Description: as for outcome 14
Time Frame: Day 30
Population: Zero participants were analyzed.
Arm/Group | IMC-1121B (Ramucirumab) + Mitoxantrone + Prednisone
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | IMC-A12 + Mitoxantrone + Prednisone | IMC-1121B (Ramucirumab) + Mitoxantrone + Prednisone
Serious Adverse Events (participants affected / at risk) | 40/66 | 36/66
Other Adverse Events (participants affected / at risk) | 65/66 | 66/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IMC-A12 + Mitoxantrone + Prednisone (N=66) | IMC-1121B (Ramucirumab) + Mitoxantrone + Prednisone (N=66)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
DISSEMINATED INTRAVASCULAR COAGULATION (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 2 (2) | 2 (2) — Event resulted in one death in IMC-1121B arm
LEUKOPENIA (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
NEUTROPENIA (Blood and lymphatic system disorders) | 2 (3) | 1 (1)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 (4) | 1 (1)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 2 (2)
CARDIAC ARREST (Cardiac disorders) | 1 (1) | 0 (0)
CARDIAC FAILURE ACUTE (Cardiac disorders) | 0 (0) | 1 (1)
HYPERTENSIVE CARDIOMYOPATHY (Cardiac disorders) | 1 (1) | 0 (0)
LEFT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 0 (0) | 2 (2)
MYOCARDIAL INFARCTION (Cardiac disorders) | 2 (2) | 0 (0)
SICK SINUS SYNDROME (Cardiac disorders) | 1 (1) | 0 (0)
RETINAL TEAR (Eye disorders) | 0 (0) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 (3) | 1 (1)
COLITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 3 (3) | 1 (1)
GASTROINTESTINAL PERFORATION (Gastrointestinal disorders) | 1 (1) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 2 (2) | 2 (3)
RECTAL PERFORATION (Gastrointestinal disorders) | 0 (0) | 1 (1)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 1 (2)
VOMITING (Gastrointestinal disorders) | 1 (1) | 2 (3)
ASTHENIA (General disorders) | 2 (2) | 0 (0)
DISEASE PROGRESSION (General disorders) | 8 (8) | 2 (2)
FATIGUE (General disorders) | 2 (2) | 0 (0)
INFUSION RELATED REACTION (General disorders) | 0 (0) | 2 (2)
PAIN (General disorders) | 1 (1) | 1 (1)
PYREXIA (General disorders) | 2 (3) | 1 (1)
ANAPHYLACTIC REACTION (Immune system disorders) | 0 (0) | 1 (1)
BACTERAEMIA (Infections and infestations) | 1 (1) | 0 (0)
CELLULITIS (Infections and infestations) | 1 (1) | 0 (0)
DIVERTICULITIS (Infections and infestations) | 0 (0) | 1 (1)
OSTEOMYELITIS (Infections and infestations) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 2 (2) | 1 (1) — Event resulted in one death in IMC-1121B arm
SEPSIS (Infections and infestations) | 1 (1) | 1 (1) — Event resulted in one death in IMC-A12 arm
SEPTIC SHOCK (Infections and infestations) | 0 (0) | 1 (1)
SOFT TISSUE INFECTION (Infections and infestations) | 1 (1) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1)
UROSEPSIS (Infections and infestations) | 0 (0) | 1 (1)
WOUND INFECTION (Infections and infestations) | 0 (0) | 1 (1)
EXPIRED DRUG ADMINISTERED (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
INCORRECT DOSE ADMINISTERED (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
MEDICATION ERROR (Injury, poisoning and procedural complications) | 0 (0) | 4 (4)
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
BLOOD CREATININE INCREASED (Investigations) | 1 (1) | 0 (0)
ANOREXIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
CACHEXIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Event resulted in death
DEHYDRATION (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
FAILURE TO THRIVE (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 (2) | 1 (1)
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
CANCER PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
METASTASES TO BONE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
METASTASES TO CENTRAL NERVOUS SYSTEM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
AUTONOMIC NEUROPATHY (Nervous system disorders) | 1 (1) | 0 (0)
CENTRAL NERVOUS SYSTEM MASS (Nervous system disorders) | 1 (1) | 0 (0)
CONVULSION (Nervous system disorders) | 0 (0) | 1 (1)
EMBOLIC STROKE (Nervous system disorders) | 0 (0) | 1 (1)
INTRAVENTRICULAR HAEMORRHAGE (Nervous system disorders) | 0 (0) | 1 (1) — Event resulted in one death in IMC-1121B arm
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 1 (1) | 0 (0)
PRESYNCOPE (Nervous system disorders) | 1 (1) | 0 (0)
SPINAL CORD COMPRESSION (Nervous system disorders) | 1 (1) | 0 (0)
SYNCOPE (Nervous system disorders) | 3 (4) | 0 (0)
TRIGEMINAL NEURALGIA (Nervous system disorders) | 0 (0) | 1 (1)
VASOGENIC CEREBRAL OEDEMA (Nervous system disorders) | 1 (1) | 0 (0)
MENTAL STATUS CHANGES (Psychiatric disorders) | 0 (0) | 1 (1)
HAEMATURIA (Renal and urinary disorders) | 2 (3) | 0 (0)
HAEMORRHAGE URINARY TRACT (Renal and urinary disorders) | 1 (1) | 0 (0)
PROTEINURIA (Renal and urinary disorders) | 1 (1) | 0 (0)
RENAL FAILURE ACUTE (Renal and urinary disorders) | 2 (2) | 1 (1)
URINARY BLADDER HAEMORRHAGE (Renal and urinary disorders) | 1 (1) | 0 (0)
URINARY RETENTION (Renal and urinary disorders) | 1 (1) | 0 (0)
TESTICULAR PAIN (Reproductive system and breast disorders) | 0 (0) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) — Events resulted in two deaths in IMC-A12 arm
DEEP VEIN THROMBOSIS (Vascular disorders) | 2 (2) | 1 (1)
HYPOTENSION (Vascular disorders) | 2 (2) | 1 (1)
PELVIC VENOUS THROMBOSIS (Vascular disorders) | 0 (0) | 1 (1)
VENA CAVA THROMBOSIS (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IMC-A12 + Mitoxantrone + Prednisone (N=66) | IMC-1121B (Ramucirumab) + Mitoxantrone + Prednisone (N=66)
ANAEMIA (Blood and lymphatic system disorders) | 23 (42) | 23 (47)
LEUKOPENIA (Blood and lymphatic system disorders) | 21 (36) | 15 (27)
LYMPHOPENIA (Blood and lymphatic system disorders) | 4 (8) | 1 (1)
NEUTROPENIA (Blood and lymphatic system disorders) | 28 (43) | 24 (43)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 12 (34) | 23 (51)
LACRIMATION INCREASED (Eye disorders) | 5 (7) | 6 (6)
ABDOMINAL PAIN (Gastrointestinal disorders) | 5 (6) | 9 (12)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 (1) | 4 (4)
CONSTIPATION (Gastrointestinal disorders) | 27 (38) | 24 (30)
DIARRHOEA (Gastrointestinal disorders) | 29 (68) | 29 (55)
DRY MOUTH (Gastrointestinal disorders) | 7 (7) | 8 (9)
DYSPEPSIA (Gastrointestinal disorders) | 8 (8) | 7 (8)
HAEMORRHOIDS (Gastrointestinal disorders) | 5 (5) | 3 (3)
NAUSEA (Gastrointestinal disorders) | 34 (55) | 31 (56)
STOMATITIS (Gastrointestinal disorders) | 7 (7) | 15 (18)
VOMITING (Gastrointestinal disorders) | 18 (24) | 19 (31)
ASTHENIA (General disorders) | 5 (5) | 12 (16)
CHILLS (General disorders) | 4 (5) | 9 (9)
FATIGUE (General disorders) | 48 (130) | 47 (97)
MUCOSAL INFLAMMATION (General disorders) | 4 (5) | 4 (4)
OEDEMA PERIPHERAL (General disorders) | 10 (13) | 14 (21)
PYREXIA (General disorders) | 10 (11) | 11 (12)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 (4) | 10 (12)
URINARY TRACT INFECTION (Infections and infestations) | 8 (9) | 4 (7)
FALL (Injury, poisoning and procedural complications) | 4 (5) | 3 (3)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 4 (4) | 7 (7)
BLOOD CREATININE INCREASED (Investigations) | 6 (13) | 2 (5)
EJECTION FRACTION DECREASED (Investigations) | 6 (8) | 11 (13)
WEIGHT DECREASED (Investigations) | 43 (94) | 40 (87)
ANOREXIA (Metabolism and nutrition disorders) | 35 (56) | 31 (45)
DEHYDRATION (Metabolism and nutrition disorders) | 15 (19) | 4 (4)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 31 (64) | 8 (15)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 4 (10) | 4 (8)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 6 (7) | 4 (5)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 4 (4) | 9 (21)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 16 (20) | 16 (29)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 13 (18) | 15 (18)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 4 (7) | 4 (5)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (4)
GROIN PAIN (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 13 (18) | 4 (4)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 7 (8) | 3 (3)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 5 (5) | 4 (4)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 9 (13) | 6 (10)
MYALGIA (Musculoskeletal and connective tissue disorders) | 5 (6) | 4 (7)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 4 (4) | 10 (21)
PAIN IN JAW (Musculoskeletal and connective tissue disorders) | 4 (7) | 2 (5)
DIZZINESS (Nervous system disorders) | 9 (13) | 12 (14)
DYSGEUSIA (Nervous system disorders) | 12 (18) | 10 (11)
HEADACHE (Nervous system disorders) | 2 (6) | 13 (18)
HYPOAESTHESIA (Nervous system disorders) | 2 (4) | 4 (4)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 2 (6) | 6 (8)
PARAESTHESIA (Nervous system disorders) | 1 (1) | 5 (5)
INSOMNIA (Psychiatric disorders) | 5 (6) | 10 (11)
CHROMATURIA (Renal and urinary disorders) | 5 (5) | 2 (2)
DYSURIA (Renal and urinary disorders) | 3 (5) | 4 (4)
NOCTURIA (Renal and urinary disorders) | 11 (12) | 5 (5)
POLLAKIURIA (Renal and urinary disorders) | 2 (2) | 4 (4)
PROTEINURIA (Renal and urinary disorders) | 3 (5) | 10 (32)
COUGH (Respiratory, thoracic and mediastinal disorders) | 13 (19) | 12 (13)
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 11 (14)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 12 (15) | 21 (28)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 11 (12)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 13 (18)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 6 (9)
PARANASAL SINUS HYPERSECRETION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
POSTNASAL DRIP (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
DRY SKIN (Skin and subcutaneous tissue disorders) | 6 (6) | 2 (2)
ECCHYMOSIS (Skin and subcutaneous tissue disorders) | 10 (11) | 16 (19)
NAIL DISORDER (Skin and subcutaneous tissue disorders) | 9 (16) | 3 (3)
HYPERTENSION (Vascular disorders) | 5 (5) | 23 (28)
HYPOTENSION (Vascular disorders) | 8 (8) | 5 (5)
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 4 (5) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators agreed to delay independently publishing or disclosing data, findings or conclusions from the study except as part of a multi-center publication. Upon study publication or if the draft publication is not produced within approximately 6 months of the final report of the study results, investigators may independently publish, subject to confidential information review/redaction by sponsor. The sponsor may request publication delay up to 90 days to seek patent protection.